CLINICAL TRIAL: NCT03441854
Title: Effects of High-Flow Nasal Cannula Versus Conventional Oxygen Therapy After Extubation in Liver Transplantation: Matched Control Study.
Brief Title: High-Flow Nasal Cannula Versus Conventional Oxygen Therapy After Extubation in Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, FERRONE GIULIANO, MD, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 1701/18
Record Dates: First submitted 2018-02-05; First posted 2018-02-22 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Gas Exchange
Keywords: Gas exchange; Non invasive ventilation; Liver transplantation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HFNC group: The investigators will prospectively include 30 patients admitted to 13- bed PICU after liver transplantation and treated with HFNC oxygen delivery after extubation.
  Interventions: Device: HFNC group
- Control Group: For each study group patient, a match control subject (matching criteria: age ± 10%, PaO2/FiO2 ± 30, diagnosis, Model for End-Stage Liver Disease (MELD) ± 10%) will be chosen from a group of 70 patients treated with conventional oxygen delivery (Venturi Mask) during the previous 2 years.

INTERVENTIONS:
Device: HFNC group — Application of HFNC oxygen delivery after extubation.
  Groups: HFNC group

SUMMARY:
Humidified oxygen therapy via high-flow nasal cannula (HFNC) is a recently available technique delivering heated and humidified high flow oxygen through simple nasal prongs. In immunocompetent patients HFNC can help generating low levels of Continuous Positive Airway Pressure (CPAP) due to the high flow of fresh gas, improving comfort and oxygenation, and it attenuates signs of respiratory distress compared with non-rebreathing oxygen face mask such as Venturi mask. Moreover, HFNC is considered to have several physiological advantages compared with other standard oxygen therapies, including the provision of positive end-expiratory pressure (PEEP), constant inspiratory oxygen fraction (FiO2), and good humidification. More importantly, it can reduce the anatomical dead space. For its advantages over conventional oxygen delivery system in patients undergoing abdominal surgery or Thoracoscopic Lobectomy, the investigators are currently and according to clinical practice using HFNC oxygen delivery in Liver transplantation after extubation, in our Post-Operative Intensive Care Unit (PICU).

Due to recipients' generally poor preoperative clinical conditions, the extensive surgical field and long operating times, post-operative respiratory disorders are very common after liver transplantation and they significantly contribute to the related morbidity and mortality, both in the acute postoperative stage and in the long term. Several factors are involved in the onset of postoperative pulmonary complications (PPCs), and many preoperative and intraoperative variables have been associated with different degrees of severity of respiratory impairment after liver transplantation. In the early stages after transplantation, pulmonary complications may prolong intubation time and increase the risk of systemic infective complications. Prolonged mechanical ventilation due to refractory respiratory failure is an extremely morbid event, as this event is a marker of poor recipient recovery, predisposes a recipient to long term ventilator dependency and predicts further complications.

In this matched control study, the investigators hypothesize that HFNC treatment might be superior to conventional oxygen therapy in terms of post-operative gas exchange and post-operative pulmonary complications for patients undergoing liver transplantation after extubation.

DETAILED DESCRIPTION:
Humidified oxygen therapy via high-flow nasal cannula (HFNC) is a recently available technique delivering heated and humidified high flow oxygen through simple nasal prongs. HFNC provides flows up to 60 L/min of heated air and oxygen at a constant fraction of inspired oxygen (FiO 2 ) up to 1.0. Several studies (1-3) have demonstrated that in immunocompetent patients HFNC can help generating low levels of CPAP due to the high flow of fresh gas, improving comfort and oxygenation, and it attenuates signs of respiratory distress compared with non-rebreathing oxygen face mask such as Venturi mask. Moreover, HFNC is considered to have several physiological advantages compared with other standard oxygen therapies, including the provision of positive end-expiratory pressure (PEEP), constant FiO2, and good humidification. More importantly, it can reduce the anatomical dead space. Several studies (1-4) demonstrated the efficacy of HFNC in reducing signs of respiratory distress compared to conventional oxygen delivery such as Venturi mask. For its advantages over conventional oxygen delivery system in patients undergoing abdominal surgery or Thoracoscopic Lobectomy (5,6), the investigators are currently and according to clinical practice using HFNC oxygen delivery in Liver transplantation after extubation, in our Post-Operative Intensive Care Unit (PICU).

Due to recipients' generally poor preoperative clinical conditions, the extensive surgical field and long operating times, post-operative respiratory disorders are very common after liver transplantation and they significantly contribute to the related morbidity and mortality, both in the acute postoperative stage and in the long term. Several factors are involved in the onset of postoperative pulmonary complications (PPCs), and many preoperative and intraoperative variables have been associated with different degrees of severity of respiratory impairment after liver transplantation (7). Although refinements in surgical techniques, antimicrobial prophylaxis, immunosuppression, anesthesia, and intensive care management have most likely altered the frequency and overall spectrum of post-liver transplantation respiratory disorders, it is still common for pulmonary infiltrates, atelectasis, pleural exudates, and other radiological abnormalities to be documented on chest X-ray at any time during a patient's stay at an intensive care unit. All of these respiratory disorders can affect lung compliance and alveolar gas exchange and, when severe, may necessitate tracheal intubation and mechanical ventilation. In the early stages after transplantation, pulmonary complications may prolong intubation time and increase the risk of systemic infective complications. Prolonged mechanical ventilation due to refractory respiratory failure is an extremely morbid event, as this event is a marker of poor recipient recovery, predisposes a recipient to long term ventilator dependency and predicts further complications.

In this patients with high risk of PPCs, the application of increased flow rates through HFNC could progressively reduce inspiratory effort and improve lung aeration, dynamic compliance and oxygenation as demonstrated in patients with acute hypoxemic respiratory failure (8).

In this matched control study, the investigators hypothesize that HFNC treatment might be superior to conventional oxygen therapy in terms of post-operative gas exchange and post-operative pulmonary complications for patients undergoing liver transplantation after extubation.

ELIGIBILITY:
Inclusion Criteria:

* Liver transplantation surgery
* Presence of criteria to start a weaning trial

Exclusion Criteria:

* Patient < 18 years
* Need of cardiovascular resuscitation
* Glasgow Coma Score ≤ 8
* Hemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: According with PICU Weaning protocol from mechanical ventilation, the investigators will be performed weaning trial and extubation after the evaluation of following conditions: 1) hemodynamic stability; 2) minimal ventilator support (pressure support ≤10 cm H2O with positive end-expiratory pressure ≤ 5 cm H2O); 3) adequate spontaneous breathing (Respiratory Rate < 25 breath.min-1).
  Successfully completed the weaning trial, the patients will be extubated and will be received humidified oxygen by HFNC at the same FiO2 as the invasive mechanical ventilation with endotracheal tube and flow rate 60 L.min
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Post- operative oxygenation | 1 hour after extubaton
  Evaluation of post-operative oxygenation measured at 1 hour after extubation

SECONDARY OUTCOMES:
Re-intubation rate | 1 week after extubaton
  Evaluation of re-intubation incidence at 1 week after extubation

CONTACTS AND LOCATIONS:
Overall Officials: Giuliano Ferrone, MD, Principal Investigator — Fondazione Policlinico Gemelli
Locations (1):
- Fondazione Policlinico Gemelli, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Corley A, Rickard CM, Aitken LM, Johnston A, Barnett A, Fraser JF, Lewis SR, Smith AF. High-flow nasal cannulae for respiratory support in adult intensive care patients. Cochrane Database Syst Rev. 2017 May 30;5(5):CD010172. doi: 10.1002/14651858.CD010172.pub2. PMID 28555461
- [Background] Mauri T, Turrini C, Eronia N, Grasselli G, Volta CA, Bellani G, Pesenti A. Physiologic Effects of High-Flow Nasal Cannula in Acute Hypoxemic Respiratory Failure. Am J Respir Crit Care Med. 2017 May 1;195(9):1207-1215. doi: 10.1164/rccm.201605-0916OC. PMID 27997805
- [Background] Futier E, Paugam-Burtz C, Godet T, Khoy-Ear L, Rozencwajg S, Delay JM, Verzilli D, Dupuis J, Chanques G, Bazin JE, Constantin JM, Pereira B, Jaber S; OPERA study investigators. Effect of early postextubation high-flow nasal cannula vs conventional oxygen therapy on hypoxaemia in patients after major abdominal surgery: a French multicentre randomised controlled trial (OPERA). Intensive Care Med. 2016 Dec;42(12):1888-1898. doi: 10.1007/s00134-016-4594-y. Epub 2016 Oct 22. PMID 27771739
- [Derived] Gaspari R, Spinazzola G, Ferrone G, Soave PM, Pintaudi G, Cutuli SL, Avolio AW, Conti G, Antonelli M. High-Flow Nasal Cannula Versus Standard Oxygen Therapy After Extubation in Liver Transplantation: A Matched Controlled Study. Respir Care. 2020 Jan;65(1):21-28. doi: 10.4187/respcare.06866. Epub 2019 Jul 3. PMID 31270177